CLINICAL TRIAL: NCT00365391
Title: Phase II Study of Bevacizumab Plus Erlotinib in Patients With Advanced Hepatocellular Cancer (HCC)
Brief Title: Bevacizumab and Erlotinib in Treating Patients With Advanced Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00136; MC044I; N01CM62205 (NIH); NCT01649076 (obsolete NCT alias)
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2013-03

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab; Erlotinib Hydrochloride

ARMS (1):
- Treatment (monoclonal antibody, enzyme inhibitor) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral erlotinib hydrochloride once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo laboratory studies to determine EGFR and phosphorylated-EGFR protein levels using initial diagnostic biopsy specimens by IHC for correlation with clinical outcome. Levels of proteins through which EGFR signals, including Akt, phosphorylated-Akt, MAPK, and phosphorylated-MAPK, are also determined using initial diagnostic biopsy specimens by IHC and correlated with clinical outcome. Total and free serum vascular endothelial growth factor levels are determined at the start of study and prior to course 3 by ELISA.
  Interventions: Biological: bevacizumab; Drug: erlotinib hydrochloride

INTERVENTIONS:
Biological: bevacizumab — Given IV, 10 mg/kg, days 1 and 15 in every cycle
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: erlotinib hydrochloride — Given orally, 150 mg, every day during each cycle.
  Other Names: CP-358,774; erlotinib; OSI-774

SUMMARY:
This phase II trial is studying how well giving bevacizumab together with erlotinib works in treating patients with advanced liver cancer. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bevacizumab and erlotinib may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving bevacizumab together with erlotinib may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the objective response rate in patients with advanced hepatocellular carcinoma treated with bevacizumab and erlotinib.

SECONDARY OBJECTIVES:

I. Evaluate the time to progression in patients treated with this regimen. II. Evaluate the overall and progression-free survival of patients treated with this regimen.

III. Evaluate the adverse events in patients treated with this regimen.

TERTIARY OBJECTIVES:

I. Determine the presence of epidermal growth factor receptor (EGFR) mutations in tumor tissue and correlate this with response rate, progression, and survival in patients treated with this regimen.

II. Evaluate the expression of molecules involved in EGFR signal transduction, including EGFR, phosphorylated-EGFR, Akt, phosphorylated-Akt, mitogen-activated protein kinase (MAPK), phosphorylated-MAPK, and HER2/neu by immunohistochemistry (from tumor tissue) and correlate these with patient outcome measures.

III. Determine the levels of vascular endothelial growth factor (VEGF) and VEGF receptors in tumor tissue as well as baseline plasma VEGF levels and correlate these with patient outcome measures.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral erlotinib hydrochloride once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo laboratory studies to determine epidermal growth factor receptor (EGFR) and phosphorylated-EGFR protein levels using initial diagnostic biopsy specimens by immunohistochemistry (IHC) for correlation with clinical outcome. Levels of proteins through which EGFR signals, including Akt, phosphorylated-Akt, mitogen-activated protein kinase (MAPK), and phosphorylated-MAPK, are also determined using initial diagnostic biopsy specimens by IHC and correlated with clinical outcome. Total and free serum vascular endothelial growth factor levels are determined at the start of study and prior to course 3 by enzyme-linked immunosorbent assays (ELISA).

After completion of study treatment, patients are followed periodically for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Absolute neutrophil count >= 1,500/mm^3
* Creatinine =< 2 mg/dL
* Albumin >= 2.5 g/dL
* Total bilirubin =< upper limit of normal (ULN)
* aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times ULN
* Alkaline phosphatase =< 5 times ULN
* Urine protein:creatinine ratio < 1.0 OR 24-hour urine protein < 1,000 mg
* Not pregnant or nursing:

No nursing for >= 6 months after completion of study treatment

* Negative pregnancy test
* Fertile patients must use effective contraception during study and for >= 6 months after completion of study treatment
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to bevacizumab or erlotinib hydrochloride
* No abnormalities of the cornea, including any of the following:

History of dry eye syndrome or Sjögren's syndrome; Congenital abnormality (e.g., Fuch's dystrophy); Abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal-Rose); Abnormal corneal sensitivity test (e.g., Schirmer test or similar tear production test)

* No stroke or transient ischemic attack within the past 6 months
* No uncontrolled high blood pressure, history of labile hypertension, or history of poor compliance with an antihypertensive regimen
* No unstable angina pectoris within the past 6 months
* No symptomatic congestive heart failure
* No myocardial infarction within the past 6 months
* No serious uncontrolled cardiac arrhythmias
* No uncontrolled diabetes mellitus
* No active or uncontrolled infection
* No impaired GI function or disease that may significantly alter the absorption of erlotinib hydrochloride (e.g., ulcerative disease, uncontrolled nausea, vomiting, or diarrhea, malabsorption syndrome, or bowel obstruction)
* Able to swallow tablets
* No psychiatric illness or social situation that would limit compliance with study requirements
* No history of nephrotic-range protein
* No history of bleeding diathesis
* No encephalopathy
* No serious nonhealing wounds, skin ulcers, or bone fractures
* No clinically significant peripheral vascular disease
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No history of a GI bleed that required procedural intervention (e.g., variceal banding, surgical shunt, transvenous intrahepatic porto-systemic shunt [TIPS]) within the past 3 months
* No significant traumatic injury within the past 28 days
* No other prior malignancy within the past 5 years except for the following:

Adequately treated basal cell or squamous cell skin cancer; Adequately treated in situ cervical cancer; Stage I or II cancer from which the patient is currently in complete remission; Stage I chronic lymphocytic leukemia

* Recovered from all therapy-related toxicities
* No more than 1 prior systemic or liver directed drug therapy including transarterial chemoembolization (TACE) (multiple TACEs will count as 1 prior regimen irrespective of their total numbers) that were used for HCC
* No chemotherapy for HCC within the past 4 weeks (6 weeks for nitrosoureas or mitomycin C)
* No biological therapy or immunotherapy for HCC within the past 4 weeks
* Prior surgery, regional therapy (e.g., transarterial embolization), liver transplantation, or other liver-directed ablative therapies of discrete lesions allowed provided any related progressive or recurrent disease is documented
* No cryotherapy, radiofrequency ablation, ethanol injection, or photodynamic therapy within the past 6 weeks:

Indicator lesions must be outside the area of prior treatment OR if the lesion is inside the area of prior treatment, there must be clear evidence of disease progression associated with that lesion

* No core biopsy within the past 7 days
* No radiotherapy within the past 4 weeks
* No prior antiangiogenesis agent or antiepidermal growth factor receptor drug
* No prior treatment with hepatic arterial infusion with chemotherapy or yttrium Y 90-labeled microspheres
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy
* Concurrent full-dose anticoagulants (e.g., warfarin) with international normalized ratio (INR) > 1.2 allowed provided the following criteria are met:

An in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant (or on a stable dose of low molecular weight heparin)

* AND (continued from above) No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels, gastrointestinal [GI] ulceration, or known varices)
* No concurrent major surgical procedures
* Histologically confirmed hepatocellular carcinoma (HCC):

  * No fibrolamellar subtype HCC
  * Advanced disease
* Not a candidate for surgical resection or liver transplantation
* Measurable disease:

  * Edges of the indicator lesion must be clearly distinct on CT scan
  * Lesions that measure at least 1 cm but less than 2 cm only must use spiral CT imaging for both pre- and post-treatment tumor assessments
* Child's Pugh classification A or B
* No primary brain tumor, brain metastasis, or other central nervous system (CNS) diseases
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Platelet count >= 75,000/mm^3
* No major surgery (e.g., laparotomy), open biopsy, or minor surgery (e.g., insertion of a vascular access device) within the past 4 weeks
* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* No abdominal fistula, GI perforation, or intra-abdominal abscess within the past 28 days
* No concurrent prophylactic hematopoietic colony-stimulating factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-08; Primary Completion 2008-08 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Philip, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Philip PA, Mahoney MR, Holen KD, Northfelt DW, Pitot HC, Picus J, Flynn PJ, Erlichman C. Phase 2 study of bevacizumab plus erlotinib in patients with advanced hepatocellular cancer. Cancer. 2012 May 1;118(9):2424-30. doi: 10.1002/cncr.26556. Epub 2011 Sep 27. PMID 21953248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2006 and March 2008, 27 patients with advanced hepatocellular carcinoma (HCC) were accrued onto the study.
Groups:
- Treatment (Bevacizumab and Erlotinib): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral erlotinib hydrochloride once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo laboratory studies to determine epidermal growth factor receptor (EGFR) and phosphorylated-EGFR protein levels using initial diagnostic biopsy specimens by immuno-histochemistry (IHC) for correlation with clinical outcome. Levels of proteins through which EGFR signals, including Akt, phosphorylated-Akt, mitogen-activated protein kinase (MAPK), and phosphorylated-MAPK, are also determined using initial diagnostic biopsy specimens by IHC and correlated with clinical outcome. Total and free serum vascular endothelial growth factor levels are determined at the start of study and prior to course 3 by ELISA.
Period: Overall Study
Arm/Group | Treatment (Bevacizumab and Erlotinib)
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Bevacizumab and Erlotinib): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral erlotinib hydrochloride once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo laboratory studies to determine EGFR and phosphorylated-EGFR protein levels using initial diagnostic biopsy specimens by IHC for correlation with clinical outcome. Levels of proteins through which EGFR signals, including Akt, phosphorylated-Akt, MAPK, and phosphorylated-MAPK, are also determined using initial diagnostic biopsy specimens by IHC and correlated with clinical outcome. Total and free serum vascular endothelial growth factor levels are determined at the start of study and prior to course 3 by ELISA.
Arm/Group | Treatment (Bevacizumab and Erlotinib)
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years]
  All Patients | 60 [36 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Confirmed Tumor Response Defined to be Either a Complete Response (CR) or Partial Response (PR).
Description: Responses to erlotinib and bevacizumab treatment were evaluated using Response Evaluation Criteria In Solid Tumors (RECIST). A Complete Response (CR) is defined as the disappearance of all target lesions. A Partial Response (PR) is defined as at least a 30% decrease in the sum of the longest diameter of target lesions taking as reference the baseline sum of the longest diameters.
Time Frame: Patients were able to continue treatment indefinitely and were evaluated every cycle until discontinued treatment.
Population: Four patients were inevaluable because they were off the study prior to first radiologic evaluation for objective response.
Measure: Number; unit: participants
Arm/Group | Treatment (Bevacizumab and Erlotinib)
Number analyzed (Participants) | 23
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 1

2. Secondary Outcome: Survival Time
Description: Survival time is defined as the time from registration to death due to any cause. Estimated using the method of Kaplan-Meier.
Time Frame: From registration to death due to any cause, patients are followed up to 3 years after treatment
Population: All 27 patients were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Bevacizumab and Erlotinib)
Number analyzed (Participants) | 27
months | 9.5 [7.1 to 17.1]

3. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from registration to documentation of disease progression. Estimated using the method of Kaplan-Meier.
Time Frame: From registration to documentation of disease progression, up to 3 years after treatment.
Population: All 27 patients were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Bevacizumab and Erlotinib)
Number analyzed (Participants) | 27
months | 3.0 [1.8 to 7.1]

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented.
Time Frame: The date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented.
Population: No patients were analyzed for this secondary outcome due to insufficient data.
Arm/Group | Treatment (Bevacizumab and Erlotinib)
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined to be the time from the date of randomization to the date at which the patient is removed from treatment due to progression, toxicity, or refusal.
Time Frame: From the date of randomization to the date at which the patient is removed from treatment due to progression, toxicity, or refusal.
Population: All 27 patients were used in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Bevacizumab and Erlotinib)
Number analyzed (Participants) | 27
months | 2.0 [1.8 to 4.6]

ADVERSE EVENTS:
Arm/Group | Treatment (Bevacizumab and Erlotinib)
Serious Adverse Events (participants affected / at risk) | 14/27
Other Adverse Events (participants affected / at risk) | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bevacizumab and Erlotinib) (N=27)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Kidney pain (Renal and urinary disorders) | 1 (1)
Renal hemorrhage (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bevacizumab and Erlotinib) (N=27)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 (6)
Eye disorder (Eye disorders) | 1 (2)
Keratitis (Eye disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 17 (44)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 3 (7)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 13 (24)
Wound infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (12)
Alkaline phosphatase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 4 (10)
Creatinine increased (Investigations) | 2 (2)
INR increased (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 2 (7)
Weight loss (Investigations) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (7)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (3)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (2)
Proteinuria (Renal and urinary disorders) | 1 (3)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (10)
Rash desquamating (Skin and subcutaneous tissue disorders) | 19 (63)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 11 (17)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less